CLINICAL TRIAL: NCT06909071
Title: Application of the Hybrid Closed-Loop Artificial Pancreas System in Neurosurgical Perioperative Hyperglycemic Patients: An Open, Randomized Controlled Trial
Brief Title: Hybrid Closed-Loop System in Neurosurgical Perioperative Hyperglycemia: An Open RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: YXLL-2025-083
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-03

CONDITIONS: T2DM Patients With Traumatic Brain Injury

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional insulin pump group (Placebo Comparator): Based on the patient's weight, the total daily insulin requirement is calculated at 0.3~0.6U/(kg*d) and distributed before meals according to the specific conditions of the patient. Continuous glucose monitoring system is used along with daily capillary blood glucose monitoring (fasting, 2 hours after breakfast, lunch, and dinner, totaling 4 times). Insulin doses are adjusted according to the patient's blood glucose level until the target blood glucose level is achieved.
  Interventions: Device: Hybrid Closed-Loop Artificial Pancreas System
- Hybrid Closed-Loop Artificial Pancreas System Group (Experimental): The open-source hybrid closed-loop artificial pancreas system, utilizing ultra-rapid-acting insulin, was employed for perioperative blood glucose management in neurosurgery. Insulin requirements were calculated based on patient weight. The system auto-adjusted basal rates according to blood glucose, while bolus treatments were manually inputted by nurses following physician instructions. Continuous and daily capillary blood glucose monitoring were conducted.
  Interventions: Device: Hybrid Closed-Loop Artificial Pancreas System

INTERVENTIONS:
Device: Hybrid Closed-Loop Artificial Pancreas System — The total daily insulin requirement is calculated as 0.3 - 0.6 U/(kg·d) according to patient's weight. The system automatically adjusts the basal rate during operation. Nurses enter bolus dose orders in AAPS software as directed by physicians. Blood glucose is monitored via continuous glucose monitoring and 4 daily fingerstick measurements (fasting and 2 hours after each meal).

SUMMARY:
In this study, we plan to use an open-source hybrid closed-loop artificial pancreas system and a combination of a traditional insulin pump and continuous glucose monitoring (CGM) respectively to conduct short-term intensive insulin treatment for patients with type 2 diabetes mellitus (T2DM) during the perioperative period who are hospitalized in the Department of Neurosurgery of Shanxi Bethune Hospital. By comparing the blood glucose control status of patients under different intensive insulin treatment regimens and other clinical indicators such as postoperative complications, we will comprehensively evaluate the clinical efficacy and safety of the hybrid closed-loop artificial pancreas system.

DETAILED DESCRIPTION:
According to the inclusion and exclusion criteria, 40 perioperative patients with type 2 diabetes mellitus (T2DM) will be screened and enrolled from the neurosurgical ward of Shanxi Bethune Hospital. They will be randomly divided into two groups: 20 patients in the hybrid closed-loop artificial pancreas system group and 20 patients in the traditional pump combined with continuous glucose monitoring (CGM) group. Both groups of patients will use continuous glucose monitoring to measure blood glucose levels. After collecting baseline data, the two groups of patients will receive short-term intensive insulin therapy according to the above-mentioned plans. Relevant clinical data will be collected during and after the treatment to compare the advantages and disadvantages of the two intensive insulin treatment plans in controlling blood glucose levels in perioperative T2DM patients undergoing neurosurgery and their impact on complications.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years old.
2. Patients who have undergone neurosurgical procedures for intracranial hemorrhage (including subdural hemorrhage, basal ganglia hemorrhage, and subarachnoid hemorrhage), have a Glasgow Coma Scale score of 12 or higher after leaving the intensive care unit, receive enteral nutrition postoperatively, and have a previously established diagnosis of type 2 diabetes mellitus, or meet the diagnostic criteria for type 2 diabetes mellitus in the "Chinese Guidelines for the Prevention and Treatment of Type 2 Diabetes" (2020 edition) .
3. Fasting blood glucose ≥ 7.0 mmol/L or random blood glucose ≥ 11.1 mmol/L.
4. Those who have signed the informed consent form and are willing to participate in this clinical trial voluntarily.

Exclusion Criteria:

1. Patients with diabetic emergencies, such as diabetic ketoacidosis, hyperglycemic hyperosmolar coma, etc.
2. Patients with type 1 diabetes or other special types of diabetes.
3. Patients with severe cardiac and renal dysfunction: those with cardiac function above grade III; those with serum creatinine exceeding 442 μmol/L.
4. Patients with diseases that affect glucose metabolism, such as hyperthyroidism, hypothyroidism, Cushing's syndrome, etc.
5. Patients who are allergic to the drugs involved in the clinical diagnosis and treatment plan.
6. Populations and contraindications that are not suitable for insulin pump treatment.
7. Patients with allergic constitution and those who are allergic to adhesive tape.
8. Patients with skin diseases such as rashes and prurigo, or those with abnormal coagulation function.
9. Patients with impaired consciousness or mental diseases, who lack self-control and cannot express themselves clearly.
10. Other situations that the researcher deems inappropriate for participating in the clinical trial.
11. Patients who develop severe complications during or after surgery and are judged by the researcher as unfit for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Time in Range (TIR) | During the 5- to 7-day period of hospitalization
  The percentage of time that blood glucose is within the target range of 6.0-12.0 mmol/L. The calculation formula is: TIR = (Time within the target range / Total time) × 100%

SECONDARY OUTCOMES:
Blood glucose target criteria | During the 5- to 7-day period of hospitalization
  FPG (fasting plasma glucose) or pre-prandial blood glucose of 8~10 mmol/L, 2hPG (2-hour postprandial glucose) or blood glucose at any time point when unable to eat is 8~12 mmol/L. General criteria: FPG or pre-prandial blood glucose of 6~8 mmol/L, 2hPG or blood glucose at any time point when unable to eat is 8~10 mmol/L (Expert Consensus on Perioperative Blood Glucose Monitoring for Adults - 2021) . The blood glucose target achievement rate within 1 week of insulin intensification therapy is calculated using the formula: Blood glucose target achievement rate = Number of patients achieving blood glucose targets / Total number of patients * 100%.
Time Below Range (TBR)、Time Above Range (TAR) | During the 5- to 7-day period of hospitalization
  Time Below Range (TBR) refers to the percentage of time when blood glucose is below the target range, that is, blood glucose < 3.9 mmol/L. The calculation formula is: TBR = (Time with blood glucose < 3.9 mmol/L) / Total Time × 100%.
  Time Above Range (TAR) refers to the percentage of time when blood glucose is above the target range, that is, blood glucose > 10.0 mmol/L. The calculation formula is: TAR = (Time with blood glucose > 10.0 mmol/L) / Total Time × 100%.
Hypoglycemia Incidence Rate | During the 5- to 7-day period of hospitalization
  Using a blood glucose range of 3.0 - 3.9 mmol/L as the diagnostic criterion for hypoglycemia, the incidence of hypoglycemia during the treatment process in the two groups was counted and compared. Taking a blood glucose level < 3.0 mmol/L as the diagnostic criterion for severe hypoglycemia, the incidence of severe hypoglycemia during the treatment process in the two groups was also counted and compared.
Blood glucose fluctuation level (IQR) | During the 5- to 7-day period of hospitalization
  The 25th and 75th percentile values of the blood glucose fluctuation range
Perioperative Infection Rate and Inflammatory Markers | During the 5- to 7-day period of hospitalization
  The percentage of patients with fever, positive bacterial culture of incision secretions, other secretions or blood during the perioperative period, calculated as (Number of patients with positive results / Total number of patients) × 100%. Perioperative inflammatory indicators include white blood cell count (WBC), percentage of neutrophils, erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), procalcitonin, etc.
Adverse event（AE）、Serious adverse event（SAE） | During the 5- to 7-day period of hospitalization
  Adverse events are defined as any unfavorable medical events that occur during the use of the investigational medical device, regardless of whether they are related to the device. Serious adverse events are defined as events that result in death or a serious deterioration of the health status during the clinical trial. The incidences of adverse events and serious adverse events during the treatment process in the three groups were statistically analyzed and compared.
Perioperative infection rate and inflammatory markers | During the 5- to 7-day period of hospitalization
  The perioperative infection rate is calculated as the number of patients who develop fever, have incision secretions, positive bacterial cultures from other secretions or blood during the perioperative period divided by the total number of patients, multiplied by 100%. Perioperative inflammatory markers include white blood cell count (WBC), percentage of neutrophils, erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), procalcitonin, etc.
Suture removal time, total hospital stay days, and postoperative hospital stay days | During the 5- to 7-day period of hospitalization
  Suture removal time, total hospital stay days, and postoperative hospital stay days

CONTACTS AND LOCATIONS:
Locations (1):
- Shanxi Bethune Hospital, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No
If there is a need to use data, please contact the person in charge and follow the relevant procedures to achieve data sharing. Without permission, do not use the data directly.